CLINICAL TRIAL: NCT03786185
Title: Neuroplasticity of Multisensory Cortical Areas Induced by Computerized Musical Training, Across the Life Span: a Translational Approach
Brief Title: Neuroplasticity of Multisensory Cortical Areas Induced by Musical Training: a Translational Approach (MusicPlast)
Acronym: MusicPlast
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Panos Bamidis, Associate Professor, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2089
Record Dates: First submitted 2018-12-20; First posted 2018-12-24 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Dyslexia; Aging Problems
Keywords: Neuroplasticity; Computerized training; Music reading; Multisensory training
MeSH Terms: conditions — Dyslexia

STUDY DESIGN:
Intervention Model Description: This is a 2x2x2 mixed model design with between subjects factors condition (congruent and incongruent) and age group (adolescent, adults, elderlies) and within subjects factor time (pre, post).
Who Masked: Participant
Masking Description: The participant is not aware of the group (intervention or control) in which s/he belongs.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Adolescents with dyslexia (Experimental): MusicPlast training
  Interventions: Behavioral: MusicPlast
- Adolescents without dyslexia (Active Comparator): MusicPlast training
  Interventions: Behavioral: MusicPlast
- Young Adults (Experimental): MusicPlast training
  Interventions: Behavioral: MusicPlast
- Young Adults Control (Active Comparator): MusicPlast Control, in a similar design as MusicPlast
  Interventions: Behavioral: MusicPlast Control
- Seniors (Experimental): MusicPlast training
  Interventions: Behavioral: MusicPlast

INTERVENTIONS:
Behavioral: MusicPlast — Each subject will receive 20 sessions of the computerized training based on a simplified music reading protocol. The training will be provided via a smartphone or a tablet. Each training session will last for 20 minutes and the log file will be directly available to the researcher, allowing him/her to follow subject's timely participation. The stimuli used in the training protocol will consist of a visual image showing a circle on top of a background of 5 horizontal lines. The auditory part of the stimulus will consist of piano melodies of known songs. The position of the circle within the five lines will either follow the rule "the higher the pitch of the tone, the higher the position of the circle" or it will violate the above rule. The task requires audiovisual integration.
  Arms: Adolescents with dyslexia; Adolescents without dyslexia; Seniors; Young Adults
Behavioral: MusicPlast Control — Each subject will receive 20 sessions of the computerized training within a period of 4 weeks, aiming to train visual search via spot-the-difference tasks and identification of dissonance in music. Auditory and visual stimuli are concurrently presented, but do not require audiovisual integration.
  Arms: Young Adults Control

SUMMARY:
Exploiting recent methodological advancements, several neuroimaging studies suggested that multisensory integration emerges from a dynamic interplay of distributed regions operating in large-scale networks. Nonetheless, the cortical structures and neuronal networks underlying the development of multisensory perception and plasticity, throughout the life span, have not yet been studied in detail. A special case of multisensory training is musical training, which utilizes stimulus' structural complexity, as well as the emotional drive that music is generating to the subjects, in order to induce augmented neuroplastic effects.

Retaining the extensive neuroplastic characteristics of music training, MUSICPLAST will develop, investigate and deliver a computer provided multisensory training protocol that aims to induce neuroplastic changes in frontotemporal cortical areas. More specifically, the goal of the proposed project is threefold: (a) The in-depth understanding and modeling of the developmental trajectory of the cortical networks underlying multisensory perception, (b) the modeling of the developmental trajectory of the cortical networks underlying multisensory plasticity throughout the life span of healthy subjects; and (c) the translation of this model in a computer provided multisensory training intervention protocol, which will cause beneficial neuroplastic changes in pathological populations. Electroencephalographic, behavioral and neuropsychological measurements, and advanced data analysis procedures, pre- and post the training application are going to be employed in order to evaluate the resulting neuroplasticity holistically. The proposed protocol will also be translated into an applied intervention for 2 groups of pathological population, for which there are strong evidence that a multisensory cognitive training based on music may provide beneficial neuroplastic changes: elderlies suffering from mild cognitive Impairment and adolescents with dyslexia.

The project is performed in the Laboratory of Medical Physics of the Aristotle University of Thessaloniki. It takes advantage of the extensive background of the laboratory in music and neuroscience, in multisensory perception and in applications that translate basic neuroscientific knowledge into computer based interventions for young adults and elderlies, building up a solid neuroscientific ground on which multidisciplinary characteristics of the project stand.

DETAILED DESCRIPTION:
Goals and research questions

The first goal of MUSICPLAST is to explore in-depth the development of audiovisual perception in the healthy human brain describing in detail the corresponding cortical networks involved. High density EEG measurements (128 channels) are going to be employed for the realization of this goal following a stimulation protocol which incorporates auditory, visual and audiovisual correspondences in a unified multisensory oddball paradigm. Behavioral and neuropsychological evaluation of the multisensory perceptual abilities of the subjects will be performed in order to achieve a holistic understanding of the phenomenon. The within subjects comparison of the different conditions will reveal the corresponding network, while the between subjects, its developmental trajectory. The hypothesis of this experiment, is that the network underlying audiovisual perception will be comprised from cortical areas connecting widespread regions including dorsolateral regions of the frontal cortex. Regarding its development, and based on the fact that behaviorally multisensory integration continues to improve in healthy aging, it is hypothesized that the network will be reorganized showing enhanced density and efficiency as the age progresses.

The second goal of MUSICPLAST is to explore in-depth the plasticity of the cortical network underlying audiovisual perception in the healthy human brain, as induced via a computer provided short-term musical reading training. Pre- and post- training high-density EEG, behavioral and neuropsychological measurements are going to be employed for the realization of this goal following the same stimulation paradigm as for the previously mentioned goal. The hypothesis of this experiment, is that the network underlying audiovisual perception will be reorganized showing enhanced global density and efficiency, greater connectivity between temporal and frontopolar regions and a gradual decline of the amount of plasticity as a result of the age increase.

The third goal of MUSICPLAST is to evaluate the effectiveness of the proposed computerized music reading training protocol as a tool that will promote beneficial neuroplastic changes in pathological populations and specifically, dyslectic adolescents and elderlies. Pre- and post- training high-density EEG, behavioral and neuropsychological measurements are going to be employed for the realization of this goal following the same stimulation paradigm as for the previously mentioned goals. The hypothesis of this experiment, is that the network underlying audiovisual perception will be beneficially reorganized due to the training showing enhanced global density and efficiency, greater connectivity between temporal and frontopolar regions and that these changes will be accompanied from improvement in the corresponding behavioral and neuropsychological evaluation.

Research design and methodology Participants

A sample size analysis was conducted via G-Power based on the data from a previous relevant study of the PI and indicated that the desired sample size in order to reach a power of 0.8 and a two sided significance level of a = 0.05 is 13 subjects in each group. In order to account for possible dropouts, MUSICPLAST will include 20 subjects in each group [adolescents (n = 20), young adults (n = 20), elderlies (n = 20) and controls (n=20)]. The study will be conducted according to the declaration of Helsinki with regard to the participation of human subjects in research.

EEG and behavioral measurements

Prior to the beginning of the training and after its completion, the participants will be subjected into 2 electroencephalographic measurements. The recordings will be performed in an electromagnetically shielded room located in the Medical Physics Laboratory of AUTH using a Nihon Kohden EEG-1200 system with 128 active electrodes. The first measurement will be of resting state activity, allowing a network analysis of resting state cortical connectivity while the second will record Event Potentials via a multisensory oddball paradigm which is appropriately adjusted for audiovisual perception, as it incorporates audiovisual, auditory and visual mismatches within one run. This paradigm has been proposed and successfully applied in a series of studies by the PI and it allows both a spatiotemporal analysis of the cortical activity as well as a functional connectivity analysis.

Concurrently to the EEG measurements the subjects will respond behaviorally via button presses to an audiovisual congruency task on which they have to evaluate whether the images presented correspond to the tones they hear based on the rule "the higher the pitch of the tone - the higher the position of the circle". This measurement will allow the behavioral evaluation of the discrimination accuracy of congruent and incongruent audiovisual stimuli.

Prior to the beginning of the training and after its completion, the participants will be subjected into a neuropsychological evaluation, which will consist of a battery including the following tests:

All subjects:

Stroop Test Trail A and B Digit Span Test Performance Subtest of Wechsler Intelligence Scale Children III or Wechsler Adult Intelligence Scale according to the age.

Elderlies only:

Mini Mental State Examination (MMSE) Montreal Cognitive Assessment (MoCA) Geriatric Depression Scale

Dyslectics only:

Word and nonword reading Word and nonword spelling Phonological ability

Intervention - MUSICPLAST training protocol

Each subject will receive 20 sessions of the computerized training based on a simplified music reading within a period of 4 weeks. The training will be provided via a smartphone or a tablet. The application will record a log file for each training session, which will last for 20 minutes and the log file will be directly available to the researcher, allowing him/her to follow the timely participation and commitment of the subject. The stimuli used in the training protocol will be constructed along the same principles of the audiovisual stimulus patterns used in the EEG recordings: a visual image will show a circle on top of a background of 5 horizontal lines. The duration of the patterns will be of a mean duration of 10 seconds.

The position of the circle within the five lines will either follow the rule "the higher the pitch of the tone, the higher the position of the circle" or it will violate the above rule. This rule was in principle followed also in previous studies conducted by the PI with positive results regarding the induced neuroplasticity. The visual images will only represent the frequency of the pitch and not the rhythmical pattern. The participant will have to respond at the end of each trial via a button press whether the audiovisual input confirmed or violated the above presented rule. A feedback image of a smiling face for the correct responses or a not smiling face for the incorrect responses will be provided for each trial. The protocol will be of adjusted difficulty, having 5 levels of difficulty which will be based on 2 different factors: the presentation speed, and the difficulty of the musical pattern. In contrast to the EEG measurement procedure, during which the melodic patterns will be unknown to the subjects, the melodic patterns used in the training will be comprised of short but identifiable parts of known musical pieces in order to engage the participants and to provoke emotional response. The training will be improved in comparison to the corresponding previous studies of the PI by providing feedback and by the use of known musical pieces which will induce an emotional response to the trainees.

EEG data analysis and statistical procedures

The EEG data collected will be pre-processed using the Brain Electrical Source Analysis software (BESA research, version 6, Megis Software, Heidelberg, Germany). The recorded data will be separated in epochs of 1000 ms including a pre-stimulus interval of 200 ms. Epochs will be baseline corrected using the interval from -100 to 0 ms. Current Density Reconstructions (CDRs) will be calculated on the neural responses of each subject and each condition using the sLORETA method55 as provided by BESA. The Matlab ® (The MathWorks, Inc., Natick, Massachusetts, United States.) toolbox HERMES56 will be used for calculating the adjacency matrix from the voxel time-series. The toolbox Network Based Statistic (NBS) will be used to statistically identify significant connections in the graphs, using a General Linear Model approach. For the statistical analysis of the data a 2 × 2 × 2 × 2 mixed model ANOVA design will be followed, with 3 within subjects factors: condition (congruent and incongruent), modality (audiovisual, auditory, and visual) and time (pre- and post- training) and one between subjects: (age group). The significance level will be set to p < 0.05 corrected for multiple comparisons via Family Wise Error correction.

ELIGIBILITY:
Group of Adolescent dyslectics

Inclusion Criteria:

* 13 - 18 years of age
* normal or corrected-to-normal hearing and vision
* Diagnosed dyslexia

Exclusion Criteria:

* any other than dyslexia, diagnosed neurological, mental, developmental or psychiatric disorder
* (ii) unrecovered neurological disorders (i.e., stroke, traumatic brain injury),
* (iii) unstable medication within the last 3 months,
* (iv) severe physical disorder, and
* (v) concurrent participation in another relevant study.

Group of Adolescent controls

Inclusion Criteria:

* 13 - 18 years of age
* normal or corrected-to-normal hearing and vision

Exclusion Criteria:

* (I) any diagnosed neurological, mental, developmental or psychiatric disorder
* (ii) unrecovered neurological disorders (i.e., stroke, traumatic brain injury),
* (iii) unstable medication within the last 3 months,
* (iv) severe physical disorder, and
* (v) concurrent participation in another relevant study.

Group of Young Adults

Inclusion Criteria:

* 18 - 35 years of age
* normal or corrected-to-normal hearing and vision

Exclusion Criteria:

* (I) any diagnosed neurological, mental, developmental or psychiatric disorder
* (ii) unrecovered neurological disorders (i.e., stroke, traumatic brain injury),
* (iii) unstable medication within the last 3 months,
* (iv) severe physical disorder, and
* (v) concurrent participation in another relevant study.

Group of Seniors

Inclusion Criteria:

* 65 - 100 years of age
* normal or corrected-to-normal hearing and vision
* normal score in a neuropsychological screening procedure which regards cognitive functionality

Exclusion Criteria:

* (i) unrecovered neurological disorders (i.e., stroke, traumatic brain injury),
* (ii) severe depression or psychological disorder,
* (iii) unstable medication within the last 3 months,
* (iv) severe physical disorder, and
* (v) concurrent participation in another relevant study.

Ages: 12 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2018-08-02 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in current density strength of the cortical activity as measured via EEG | 1 month
  Changes in cortical activity strength caused via the training. Change is defined as statistical significance in the t-test comparison of the current density strength as reconstructed via Low Resolution Electromagnetic Tomography (LORETA) algorithm on the basis of high density EEG recordings, before compared to after the training
Change in cortical connectivity as measured via EEG | 1 month
  Changes in cortical connectivity caused via the training. Change is defined as statistical significance in the t-test comparison of the Transfer Entropy estimated from the cortical activity, as reconstructed via LORETA algorithm on the basis of high density EEG recordings, before compared to after the training.

SECONDARY OUTCOMES:
Change in audiovisual integration functionality | 1 month
  Change of accuracy in the behavioral measurement testing audiovisual integration. Change is defined as statistical significance in the t-test comparison before compared to after the training.
Change in cognitive functionality | 1 month
  Change of scoring in neuropsychological tests related with attention, memory and performance. Change is defined as statistical significance in the t-test comparison before compared to after the training.

CONTACTS AND LOCATIONS:
Overall Officials: Evangelos Paraskevopoulos, PhD, Principal Investigator — Research Associate
Locations (1):
- Laboratory of Medical Physics, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: Undecided
Individual Participant Data (IPD) will be available upon the completion of the study via personal communication. Data shared will include EEG measurements, score on behavioral and psychometric data.

REFERENCES:
- [Background] Paraskevopoulos E, Kraneburg A, Herholz SC, Bamidis PD, Pantev C. Musical expertise is related to altered functional connectivity during audiovisual integration. Proc Natl Acad Sci U S A. 2015 Oct 6;112(40):12522-7. doi: 10.1073/pnas.1510662112. Epub 2015 Sep 14. PMID 26371305
- [Background] Paraskevopoulos E, Kuchenbuch A, Herholz SC, Pantev C. Multisensory integration during short-term music reading training enhances both uni- and multisensory cortical processing. J Cogn Neurosci. 2014 Oct;26(10):2224-38. doi: 10.1162/jocn_a_00620. Epub 2014 Mar 26. PMID 24669793
- [Background] Paraskevopoulos E, Kuchenbuch A, Herholz SC, Pantev C. Musical expertise induces audiovisual integration of abstract congruency rules. J Neurosci. 2012 Dec 12;32(50):18196-203. doi: 10.1523/JNEUROSCI.1947-12.2012. PMID 23238733
- See also: project web-site — https://users.auth.gr/parasvag/MusicPlast/